CLINICAL TRIAL: NCT02605213
Title: Evaluation of Effectiveness and Safety of Oral Vancomycin in Treatment of Primary Sclerosing Cholangitis.
Brief Title: Effect and Safety of Oral Vancomycin in Primary Sclerosing Cholangitis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nasser Ebrahim Daryani, Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9311366004
Record Dates: First submitted 2015-10-31; First posted 2015-11-16 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-11

CONDITIONS: Primary Sclerosing Cholangitis
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vancomycin (Experimental): Vancomyicn 250 mg every 6 hours for 12 weeks
  Interventions: Drug: Vancomycin
- Placebo (Placebo Comparator): placebo every 6 hours for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vancomycin — Vancomycin for treatment of primary sclerosing cholangitis
  Other Names: Vancomycin hydrochloride,
  Arms: Vancomycin
Drug: Placebo — Placebo for control Group of primary sclerosing vhlangitis
  Arms: Placebo

SUMMARY:
Primary sclerotic cholangitis (PSC) is an inflammatory process of sclerotic cholangitis that involves intra and extra hepatic biliary system. There is no curative treatment for this disorder. Supportive and conservative treatments are the most common therapies that used for this disease. Although treatments such as ursodeoxycholic acid (UDCA) are recommended in some situations but whereas a hypothesis is stimulatory effect of intestinal anaerobic bacteria such as cholestridium difficile as pathogenesıs of PSC, so use of antibiotics is recommended for treatment of these patients. Therefore according to the great role of anaerobic bacteria such as cholestridium difficile in pathogenesis, antibiotics such as metronidazole and vancomycin can be counted as recommended therapies in PSC. In addition some studies correlated this effect of vancomycin to its immunomudulatory effect the cause reduction of inflammation in biliary system. But with all this detail there is no finality about effectiveness of antibiotic therapy and accordingly in this study the investigators compare oral vancomycin effect versus placebo in primary sclerosing cholangitis patients.

In this double blind clinical trial 30 primary sclerosing cholangitis patients that divided in two 15 persosns group with Block Randomization method. in this study one group receive 250 mg oral vancomycin every 6 hours and other group receive placebo.

The study duration is 12 weeks . The baseline laboratory tests and 1 month and 3 months after treatment concept of; Alkaline phosphatase, ALT, AST, GGT and serum total bilirubin and clinical manifestations such as tiredness, itching and probable adverse effects such as hypotension accompanied by flushing,erythematous rash on face and upper body (red neck or red man syndrome), chills and drug fever, eosinophilia and reversible neutropenia.

ELIGIBILITY:
Inclusion Criteria:

1. primary sclerosing chollangitis diagnosis more than 3 months
2. inflammatory bowel disease with cholestasis diagnosis more than 3 months
3. confirmed RCPM
4. confirmed pathology of inflammatory bowel disease

Exclusion Criteria:

1. signs of uncompensated cirrhosis like: hepatic encephalopathy, esophageal varices bleeding
2. gastrointestinal cancer or hepatic cancer
3. immunosuppressive agent using for hepatic problem (not vancomycine hypersensitivity)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
comparison of laboratory data Alkalyne phosphatase between baseline and after treatment | 12 weeks
  Alkaline phosphatase
comparison of laboratory data ALT between baseline and after treatment | 12 weeks
  ALT
comparison of laboratory data AST between baseline and after treatment | 12 weeks
  AST
comparison of laboratory data GGT between baseline and after treatment | 12 weeks
  GGT
comparison of laboratory data serum total bilirubin between baseline and after treatment | 12 weeks
  serum total bilirubin
baseline data | baseline
  serum Albumin

SECONDARY OUTCOMES:
Number of participants with adverse events | 12 weeks
  clinical manifestations such as tiredness, itching and probable adverse effects such as hypotension accompanied by flushing,erythematous rash on face and upper body (red neck or red man syndrome), chills and drug fever, eosinophilia and reversible neutropenia.

CONTACTS AND LOCATIONS:
Overall Officials: Shahab Rahimpour, fellowship, Principal Investigator — Tehran University of Medical Sciences; Mohammad Kazem NouriTaromlou, M.D., Study Director — Tehran UMS; Naser Ebrahimi Daryani, Professor, Study Director — Tehran University of Medical Sciences; Sanam Javidanbardan, M.D., Study Director — Tehran University of Medical Sciences; Zahra Azizi, M.D., Study Director — Tehran University of Medical Sciences; Mohsen Nasiri Toosi, Professor, Study Director — Tehran University of Medical Sciences
Locations (1):
- Imam khomeini Hospital Complex, Tehran, Tehran Province, Iran